CLINICAL TRIAL: NCT01710709
Title: A 52-week, Multicenter, Open-label Study to Evaluate the Effectiveness of an Intramuscular Depot Formulation of Aripiprazole (OPC-14597) as Maintenance Treatment in Patients With Bipolar I Disorder
Brief Title: Open-label Study to Evaluate the Effectiveness of an Intramuscular Formulation of Aripiprazole (OPC-14597) as Maintenance Treatment in Patients With Bipolar I Disorder
Acronym: ATLAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-08-252
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Bipolar I
Keywords: Aripiprazole, Intramuscular (IM) Depot, Bipolar
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Aripiprazole, Intramuscular (IM) Depot
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — 400mg or 300mg, intramuscular injections every 4 weeks.

SUMMARY:
This will be an open-label uncontrolled trial to evaluate the safety and tolerability of aripiprazole IM depot administered every 4 weeks for up to 52 weeks to patients with bipolar I disorder. The trial will enroll subjects who completed Trial 31-08-250 and de novo subjects not participating in Trial 31-08-250.

DETAILED DESCRIPTION:
This will be an open-label, uncontrolled study which will enroll subjects completing Study 31-08-250 and new subjects. The treatment history of subjects prior to enrollment in the open-label study will vary according to the design of the pivotal double-blind study (i.e 31-08-250).

This open-label study will be comprised of phases similar to the pivotal double-blind study (i.e. Study 250): a screening phase (if applicable), a conversion phase (Phase A, if applicable), an oral stabilization phase (Phase B, if applicable), and an IM depot open-label maintenance phase (Phase C). Phase C will be a minimum of 28 weeks up to a 52-week treatment period with a 4 week follow up period.

During Phase C (the open-label maintenance phase) rescue medication will be allowed for subjects who do not meet stability criteria. This analysis focuses on Phase C due to ClinicalTrials.gov system limitations.

ELIGIBILITY:
Inclusion Criteria:

* Completed participation in Trial 31-08-250
* De novo subjects not participating in Trial 31-08-250
* Subjects who are able to provide written informed consent.
* Male and female subjects 18 years of age or older at time of informed consent
* Subjects who, in the investigator's judgment, require chronic treatment with an antipsychotic medication for their bipolar I disorder and would benefit from extended treatment with a long-acting injectable formulation
* Subjects who have a recurrence of mood episode or exacerbations of mood symptoms when they are not receiving treatment for their bipolar I disorder or are noncompliant with treatment for their bipolar I disorder
* Have an outpatient status

Exclusion Criteria:

* Experienced 9 or more mood episodes within the past year
* A current manic episode with a duration of > 2 years
* Currently meet DSM-IV-TR criteria for substance abuse or substance dependence; this includes the abuse of alcohol and benzodiazepines, but excludes the use of caffeine and/or nicotine
* Hypothyroidism or hyperthyroidism, unless condition has been stabilized
* Diagnosed with epilepsy or a history of seizures
* Known to be allergic, intolerant, or unresponsive to prior treatment with aripiprazole or other quinolinones
* Sexually active women of childbearing potential and sexually active men who will not commit to utilizing 2 of the approved birth control methods or who will not remain abstinent during this trial and for 180 days following the last dose of trial medication
* Females breastfeeding or pregnant (positive blood pregnancy test prior to receiving trial drug)
* Risk of committing suicide
* Abnormal laboratory test results, vital signs and ECG results
* Participated in any clinical trial other than Trial 250 with an investigational agent within the 30 days prior to screening
* Had electroconvulsive therapy (ECT) treatment during the current episode or within 3 months
* Subjects who have not met criteria for stabilization for 4 consecutive weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2012-11; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Amatniek, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc. (OPDC)
Locations (111):
- United States (65):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Rogers, Arkansas
  - Bellflower, California
  - Beverly Hills, California
  - Costa Mesa, California
  - Culver City, California
  - Garden Grove, California
  - Lemon Grove, California
  - Oakland, California
  - Orange, California
  - Pico Rivera, California
  - Riverside, California
  - San Diego, California
  - Temecula, California
  - Upland, California
  - Wildomar, California
  - Colorado Springs, Colorado
  - Gainesville, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Leesburg, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Smyrna, Georgia
  - Chicago, Illinois
  - Hinsdale, Illinois
  - Naperville, Illinois
  - Schaumburg, Illinois
  - Prairie Village, Kansas
  - Lake Charles, Louisiana
  - Baltimore, Maryland
  - Gaithersburg, Maryland
  - Boston, Massachusetts
  - O'Fallon, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Berlin, New Jersey
  - Cherry Hill, New Jersey
  - Brooklyn, New York
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Media, Pennsylvania
  - Columbia, South Carolina
  - Memphis, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Dallas, Texas
  - Plano, Texas
  - Sugar Land, Texas
  - Wichita Falls, Texas
  - Orem, Utah
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Bellevue, Washington
  - Spokane, Washington
  - Middleton, Wisconsin
- Canada (2):
  - Kentville, Nova Scotia
  - Chatham, Ontario
- France (4):
  - Élancourt
  - Limoges
  - Nîmes
  - Toulouse
- Hungary (3):
  - Budapest
  - Nyireghaza
  - Vác
- Japan (19):
  - Fukuoka
  - Fukushima
  - Gunma
  - Ibaraki
  - Iizuka
  - Kanagawa
  - Kochi
  - Kouchi
  - Kumamoto
  - Nagano-ken
  - Okayama
  - Okinawa
  - Osaka
  - Ōsaka
  - Sapporo
  - Shizuoka
  - Tokyo
  - Yamagata
  - Yatsushiro
- Malaysia (3):
  - Johor Bahru
  - Perak
  - Sarawak
- Poland (7):
  - Bydgoszcz
  - Chełmno
  - Choroszcz
  - Gdansk
  - Lublin
  - Pruszków
  - Tuszyn
- Romania (4):
  - Bucharest
  - Iași
  - Târgovişte
  - Târgu Mureş
- South Korea (3):
  - Goyang-si
  - Jeju City
  - Seoul
- Taipei, Taiwan

REFERENCES:
- [Derived] Calabrese JR, Jin N, Johnson B, Such P, Baker RA, Madera J, Hertel P, Ottinger J, Amatniek J, Kawasaki H. Aripiprazole once-monthly as maintenance treatment for bipolar I disorder: a 52-week, multicenter, open-label study. Int J Bipolar Disord. 2018 Jun 10;6(1):14. doi: 10.1186/s40345-018-0122-z. PMID 29886522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label, single-arm, uncontrolled trial evaluated aripiprazole intramuscular (IM) depot as maintenance treatment for participants with bipolar I disorder. Enrolled participants included those who had completed Trial 31-08-250 (NCT01567527) as well as de novo participants who had not participated in Trial 31-08-250.
Pre-assignment Details: Screening period was from Day -42 to Day -2. Participants from the Trial 31-08-250 entered directly into the IM Depot Maintenance Phase of Trial 31-08-252. For de novo participants, this trial consisted of Phases A-C (Conversion Phase, Oral Stabilization Phase, and IM Depot Maintenance Phase).
Groups:
- Phase C: Open-Label IM Depot Maintenance Phase: All de novo participants received open-label aripiprazole 400/300 mg IM depot and the participants who completed Trial 31-08-250 entered phase C on aripiprazole IM depot 400 mg, regardless of their last dose of IM depot. Aripiprazole IM depot injections were administered every 4 weeks for a maximum of 52 weeks. De novo participants also received daily supplemental oral aripiprazole (10 to 20 mg daily for non-Japanese sites; 6 to 18 mg for Japanese sites) for the first 2 weeks to maintain therapeutic plasma concentrations. Note: Data for Open-label aripiprazole IM depot maintenance phase (Phase C) is presented in the table below which included both rollover participants (those who had completed Trial 31-08-250 and entered into the Open-label aripiprazole IM depot maintenance phase directly) and de novo participants (ie, those who did not participate in Trial 31-08-250 and went through Screening phase, Conversion Phase, and Oral aripiprazole stabilization phase).
Period: Overall Study
Arm/Group | Phase C: Open-Label IM Depot Maintenance Phase
Started | 464
Completed | 291
Not Completed | 173
Not completed — Lost to Follow-up | 29
Not completed — Adverse Event | 48
Not completed — Participant met withdrawal criteria | 33
Not completed — Participant withdrawn by investigator | 2
Not completed — Withdrawal by Subject | 53
Not completed — Protocol Violation | 5
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Groups:
- Phase C: Open-label IM Depot Maintenance Phase: All de novo participants received open-label aripiprazole 400/300 mg IM depot and the participants who completed Trial 31-08-250 entered phase C on aripiprazole IM depot 400 mg, regardless of their last dose of IM depot. Aripiprazole IM depot injections were administered every 4 weeks for a maximum of 52 weeks. Flexible dosing with aripiprazole IM depot 300 mg and 400 mg was permitted as often as necessary during the open-label treatment period. De novo participants also received daily supplemental oral aripiprazole (10 to 20 mg daily for non-Japanese sites; 6 to 18 mg for Japanese sites) for the first 2 weeks to maintain therapeutic plasma concentrations. For participants who completed Trial 31-08-250 (some of whom had received double-blind placebo), the use of supplemental oral aripiprazole for the first ≤ 2 weeks was at the investigator's discretion based on the clinical status of the participant.
Arm/Group | Phase C: Open-label IM Depot Maintenance Phase
Number analyzed (Participants) | 464
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 458
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 268
  Male | 196
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3
  South Korea | 6
  Romania | 10
  Hungary | 4
  United States | 322
  Japan | 75
  Taiwan | 1
  Poland | 28
  Malaysia | 10
  France | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or participant enrolled in the clinical trial and which does not necessarily have to have a causal relationship with the investigational medicinal product (IMP). AEs were assessed as a criteria for safety and tolerability.
Time Frame: Up to Week 52
Population: IM Depot Maintenance Phase Safety Sample: All participants who received at least 1 dose of aripiprazole IM depot in the IM Depot Maintenance Phase. TEAEs = Treatment-emergent adverse events. discount. = discontinued (used in the table below)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase C: Open-label IM Depot Maintenance Phase
Number analyzed (Participants) | 464
Participants
  Participants with adverse events | 374
  Participants with TEAEs | 374
  Participants with serious TEAEs | 30
  Participants with severe TEAEs | 41
  Participants discontinued from IMP due to AEs | 47
  Participants discont. from IMP due to AEs or death | 48
  Deaths | 1

2. Primary Outcome: Injection Site Pain Measured by the Visual Analog Scale (VAS)
Description: Injection-site pain was evaluated by mean visual analog scale (VAS) scores as reported by the participant after each injection at visits where an injection occurred. Ratings ranged from 0 (no pain) to 100 (unbearably painful).
Time Frame: Up to Week 52
Population: All participants who received at least one dose of aripiprazole IM depot in Phase C. It is equivalent to safety set (SAF) for Phase C.
  Number analyzed = Total number of participants with at least one observation of the given parameter.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Phase C: Open-label IM Depot Maintenance Phase
Number analyzed (Participants) | 464
Units on a scale
  1ST Injection: number analyzed (Participants) | 462
  1ST Injection | 4.9 (10.7)
  2ND Injection: number analyzed (Participants) | 435
  2ND Injection | 4.1 (8.4)
  3RD Injection: number analyzed (Participants) | 422
  3RD Injection | 3.4 (7.5)
  4TH Injection: number analyzed (Participants) | 402
  4TH Injection | 3.6 (8.6)
  5TH Injection: number analyzed (Participants) | 387
  5TH Injection | 2.9 (7.9)
  6TH Injection: number analyzed (Participants) | 366
  6TH Injection | 2.4 (5.8)
  7TH Injection: number analyzed (Participants) | 353
  7TH Injection | 2.6 (7.0)
  8TH Injection: number analyzed (Participants) | 293
  8TH Injection | 2.4 (4.9)
  9TH Injection: number analyzed (Participants) | 284
  9TH Injection | 2.6 (6.6)
  10TH Injection: number analyzed (Participants) | 264
  10TH Injection | 2.5 (7.5)
  11TH Injection: number analyzed (Participants) | 255
  11TH Injection | 2.4 (6.3)
  12TH Injection: number analyzed (Participants) | 247
  12TH Injection | 1.8 (4.3)
  13TH Injection: number analyzed (Participants) | 223
  13TH Injection | 2.2 (5.5)
  Last Injection: number analyzed (Participants) | 463
  Last Injection | 2.4 (5.9)

3. Primary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Test Results
Description: Standard safety variables to be analyzed included clinical laboratory tests. Incidence of treatment emergent adverse events (TEAEs) of potential clinical relevance included abnormal values in serum chemistry, hematology, urinalysis, and other laboratory test that were identified based on pre-defined criteria. Abnormal laboratory values in participants were reported as serious adverse event/adverse events (SAE/AEs) and are reported in the SAE/other AE section of this report.
Time Frame: Up to Week 52
Population: IM Depot Maintenance Phase Safety Sample: All participants who received at least 1 dose of aripiprazole IM depot in the IM Depot Maintenance Phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase C: Open-label IM Depot Maintenance Phase
Number analyzed (Participants) | 464
Participants
  Fasting cholesterol | 53
  Fasting glucose | 39
  Fasting low-density lipoprotein cholesterol | 32
  Fasting triglycerides | 124

4. Primary Outcome: Number of Participants With Clinically Significant Abnormal Vital Signs
Description: TEAEs of potential clinical relevance included abnormal values in body weight, systolic and diastolic blood pressure, heart rate, and body temperature that were identified based on pre-defined criteria. Abnormal laboratory values in participants were reported as SAE/AEs and are reported in the SAE/other AE section of this report.
Time Frame: Up to Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase C: Open-label IM Depot Maintenance Phase
Number analyzed (Participants) | 464
Participants
  Weight gain of ≥ 7%: number analyzed (Participants) | 454
  Weight gain of ≥ 7% | 93
  Weight loss of ≥ 7%: number analyzed (Participants) | 454
  Weight loss of ≥ 7% | 66
  Blood pressure increased | 4
  Heart rate increased | 3
  Blood pressure decreased | 2
  Body temperature | 0

5. Primary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECGs)
Description: Twelve-lead ECGs were recorded at specified visits. For each time point, three 12-lead ECG recordings were obtained approximately 5 minutes apart. Additional 12-lead ECGs were permitted to be obtained at the investigator's discretion and were to always be obtained in the event of an early termination. The ECGs were evaluated at the investigational site to determine the participant's eligibility and to monitor safety during the trial.
Time Frame: Up to Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase C: Open-label IM Depot Maintenance Phase
Number analyzed (Participants) | 464
Participants
  Symmetrical T-wave inversion: number analyzed (Participants) | 412
  Symmetrical T-wave inversion | 9
  Supraventricular premature beat: number analyzed (Participants) | 412
  Supraventricular premature beat | 8
  Ventricular premature beat: number analyzed (Participants) | 412
  Ventricular premature beat | 4
  Myocardial ischemia: number analyzed (Participants) | 412
  Myocardial ischemia | 2

6. Primary Outcome: Extrapyramidal Symptoms Will be Assessed by Mean Change From Baseline on Abnormal Involuntary Movement Scale(AIMS), Simpson-Angus Scale (SAS), Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS Only Used in Japan) and Barnes Akathisia Rating Scale (BARS)
Description: AIMS: 10 items described dyskinesia signs; 0-absence/no awareness; 4-severe condition/severe distress. Total score for Items 1-10 ranges from 0 to 40; a higher score reflects severe condition. SAS:Consisted of 10 parkinsonism signs;1-no symptoms;5-severe.Total score for Items 1-10 ranges from 1 to 50;a higher score reflects severe condition.DIEPSS:A 9-item rating scale (8 assessed individual symptoms [4 categories of parkinsonism, akathisia, dystonia & dyskinesia]+1 assessed general severity) was used;0-no symptoms/normal, 4-severe.Total score (8 individual symptom items) was in range of 0 to 32 (a higher score reflects severe condition).BARS:Consisted of 4 items related to akathisia:objective observation, subjective feelings of restlessness, distress, global clinical evaluation.Only BARS global clinical assessment score has been presented and rated using scale:0-absence of symptoms;5-severe akathisia.Total BARS global score ranges from 0 to 5,a higher score reflects severe condition.
Time Frame: Baseline, Week 28, and Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Phase C: Open-label IM Depot Maintenance Phase: All de novo participants received open-label aripiprazole 400/300 mg IM depot and the participants who completed Trial 31-08-250 entered phase C on aripiprazole IM depot 400 mg, regardless of their last dose of IM depot. Aripiprazole IM depot injections were administered every 4 weeks for a maximum of 52 weeks. Flexible dosing with aripiprazole IM depot 300 mg and 400 mg was permitted as often as necessary during the open-label treatment period. De novo participants also received daily supplemental oral aripiprazole (10 to 20 mg daily for non-Japanese sites; 6 to 18 mg for Japanese sites) for the first 2 weeks to maintain therapeutic plasma concentrations. For participants who completed Trial 31-08-250 (some of whom had received double-blind placebo), the use of supplemental oral aripiprazole for the first ≤ 2 weeks was at the investigator's discretion based on the clinical status of the participant. Results using last observation carried forward (LOCF) were presented.
Arm/Group | Phase C: Open-label IM Depot Maintenance Phase
Number analyzed (Participants) | 464
Units on a scale
  AIMS, Week 28: number analyzed (Participants) | 457
  AIMS, Week 28 | 0.07 (1.00)
  AIMS, Week 52: number analyzed (Participants) | 457
  AIMS, Week 52 | 0.05 (0.97)
  SAS, Week 28: number analyzed (Participants) | 377
  SAS, Week 28 | 0.21 (1.59)
  SAS, Week 52: number analyzed (Participants) | 377
  SAS, Week 52 | 0.20 (1.58)
  DIEPSS, Week 28: number analyzed (Participants) | 75
  DIEPSS, Week 28 | 0.32 (1.29)
  DIEPSS, Week 52: number analyzed (Participants) | 75
  DIEPSS, Week 52 | 0.21 (1.11)
  BARS, Week 28: number analyzed (Participants) | 457
  BARS, Week 28 | 0.05 (0.61)
  BARS, Week 52: number analyzed (Participants) | 457
  BARS, Week 52 | 0.04 (0.60)

7. Primary Outcome: Number of Participants Experiencing Suicidal Events and Their Classification According to the Completion of Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Suicidality was monitored throughout the trial using the C-SSRS at every visit. The C-SSRS scale consisted of a screening/baseline evaluation that assessed the participant's lifetime experience and experience over the last 90 days with suicide events and suicidal ideation and a post-baseline/ "Since Last Visit" evaluation that focused on suicidality since the last trial visit.
Time Frame: Up to Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase C: Open-label IM Depot Maintenance Phase
Number analyzed (Participants) | 464
Participants
  Completed Suicide: number analyzed (Participants) | 463
  Completed Suicide | 0
  Suicide Attempt: number analyzed (Participants) | 463
  Suicide Attempt | 3
  Preparatory action toward imminent suicide: number analyzed (Participants) | 463
  Preparatory action toward imminent suicide | 4
  Suicidal ideation: number analyzed (Participants) | 463
  Suicidal ideation | 46
  Non-suicidal self-injurious behavior: number analyzed (Participants) | 463
  Non-suicidal self-injurious behavior | 4

8. Primary Outcome: Number of Participants With Injection Site Evaluations (Pain, Redness, Swelling, Induration) Measured by Investigator Rating
Description: Injection-site reactions were assessed by the investigator (or qualified designee) and the participant. Investigators rated localized pain, redness, swelling, and induration at the most recent injection site using a 4-point categorical scale (absent, mild, moderate, severe) . The participant indicated the degree of pain at the most recent injection site using a VAS. Ratings ranged from 0 (no pain) to 100 (unbearably painful). Ratings included were: 0 = absent, 1 = mild, 2 = moderate, 3 = severe. These assessments occurred at trial visits where injections occurred (scheduled and unscheduled), beginning with the first dose of open-label aripiprazole IM depot administered at the final visit of the Oral Stabilization Phase and continued through the last injection prior to the end of the IM Depot Maintenance Phase/Early termination (ET) visit (ie, evaluations were not done at end of the IM Depot Maintenance Phase/ET visit).
Time Frame: Up to Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase C: Open-label IM Depot Maintenance Phase
Number analyzed (Participants) | 464
Participants
  Injection Site Bruising | 2
  Injection Site Erythema | 1
  Injection Site Induration | 1
  Injection Site Mass | 2
  Injection Site Pain | 34
  Injection Site Swelling | 4

9. Secondary Outcome: Percentage of Participants Who Remained Stable at End of Treatment in Phase C
Description: The secondary objective was to evaluate the efficacy, as measured by the percentage of stable participants at baseline who remained stable at the end of treatment in the IM depot maintenance phase, of aripiprazole IM depot administered every 4 weeks for up to 52 weeks to subjects with bipolar I disorder.
Time Frame: Up to Week 52
Population: IM Depot Maintenance Phase Efficacy Sample: All participants who entered the IM Depot Maintenance Phase, received at least 1 dose of aripiprazole IM depot, and had at least 1 post-baseline efficacy evaluation in the IM Depot Maintenance Phase. Number analyzed is the number of participants evaluated at the specified trial week.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase C: Open-label IM Depot Maintenance Phase
Number analyzed (Participants) | 464
Percentage of participants
  Baseline: number analyzed (Participants) | 463
  Baseline | 100.00
  Week 2: number analyzed (Participants) | 430
  Week 2 | 96.98
  Week 4: number analyzed (Participants) | 432
  Week 4 | 97.22
  Week 8: number analyzed (Participants) | 413
  Week 8 | 95.64
  Week 12: number analyzed (Participants) | 406
  Week 12 | 96.31
  Week 16: number analyzed (Participants) | 396
  Week 16 | 96.46
  Week 20: number analyzed (Participants) | 381
  Week 20 | 95.54
  Week 24: number analyzed (Participants) | 361
  Week 24 | 96.40
  Week 28: number analyzed (Participants) | 346
  Week 28 | 95.09
  Week 32: number analyzed (Participants) | 287
  Week 32 | 97.91
  Week 36: number analyzed (Participants) | 271
  Week 36 | 95.94
  Week 40: number analyzed (Participants) | 255
  Week 40 | 98.04
  Week 44: number analyzed (Participants) | 249
  Week 44 | 97.59
  Week 48: number analyzed (Participants) | 243
  Week 48 | 97.53
  Week 52: number analyzed (Participants) | 237
  Week 52 | 95.78
  Last Visit: number analyzed (Participants) | 460
  Last Visit | 88.91

ADVERSE EVENTS:
Time Frame: Phase C week 1 to week 52/early termination.
Description: All participants who had received at least one dose of aripiprazole IM depot were included in safety analysis.
Arm/Group | Phase C: Open-Label IM Depot Maintenance Phase
All-Cause Mortality (participants affected / at risk) | 1/464
Serious Adverse Events (participants affected / at risk) | 30/464
Other Adverse Events (participants affected / at risk) | 367/464
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase C: Open-Label IM Depot Maintenance Phase (N=464)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Prinzmetal Angina (Cardiac disorders) | 1 (3)
Hyperprolactinaemia (Endocrine disorders) | 1 (1)
Chest Pain (General disorders) | 2 (2)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Tardive Dyskinesia (Nervous system disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (2)
Bipolar Disorder (Psychiatric disorders) | 2 (2)
Bipolar I Disorder (Psychiatric disorders) | 4 (4)
Major Depression (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 3 (3)
Social Avoidant Behaviour (Psychiatric disorders) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 4 (4)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase C: Open-Label IM Depot Maintenance Phase (N=464)
Injection site pain (General disorders) | 34 (50)
Nasopharyngitis (Infections and infestations) | 56 (87)
Upper respiratory tract infection (Infections and infestations) | 24 (27)
Weight increased (Investigations) | 62 (66)
Akathisia (Nervous system disorders) | 68 (79)
Headache (Nervous system disorders) | 29 (37)
Tremor (Nervous system disorders) | 28 (38)
Anxiety (Psychiatric disorders) | 46 (60)
Depression (Psychiatric disorders) | 26 (35)
Insomnia (Psychiatric disorders) | 51 (54)
Restlessness (Psychiatric disorders) | 23 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other